CLINICAL TRIAL: NCT06803823
Title: A Phase 2a, Multicenter, Placebo-controlled, Randomized, Double-blind, Parallel-group Study to Evaluate the Efficacy and Safety of ONO-2020 in Patients With Agitation Associated With Alzheimer's Disease Dementia
Brief Title: A Study of ONO-2020 in Patients With Agitation Associated With Alzheimer's Disease Dementia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ONO-2020-03; jRCT2041230153 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Agitation Associated With Alzheimer's Disease Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ONO-2020 (Experimental)
  Interventions: Drug: ONO-2020
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ONO-2020 — ONO-2020 group: Two ONO-2020 tablets will be orally administered once daily.
  Arms: ONO-2020
Drug: Placebo — Two ONO-2020 placebo tablets will be orally administered once daily
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of ONO-2020 in patients with agitation associated with Alzheimer's Disease dementia in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable AD according to the diagnostic criteria for AD dementia (NIA-AA 2011)
* Mini-Mental State Examination (MMSE) score ≥ 5 to ≤ 22 at the start of the treatment period
* Symptoms of agitation defined by the IPA from at least 14 days before the start of the screening period
* Neuropsychiatric Inventory-Nursing Home version (NPI-NH) Agitation/Aggression domain (NPI-NH-A/A) score ≥ 4 at the start of the treatment period.
* Patients who can participate in the study under hospitalization from 21 days before the start of the treatment period to throughout the treatment period

Exclusion Criteria:

* Diagnosis of dementia not due to AD or any other disorder with memory impairment, such as mixed dementia, vascular dementia, Lewy body dementia, dementia associated with Parkinson's disease, frontotemporal dementia, drug-induced dementia, dementia associated with human immunodeficiency virus (HIV) infection, traumatic brain injury, normal pressure hydrocephalus, or other non-AD dementia
* Any MRI or CT scan of the brain performed after the onset of dementia with findings consistent with clinically relevant CNS disease other than AD, such as vascular changes (eg, cortical cerebral infarction, multiple cerebral infarctions), space-occupying lesions (eg, tumors), or any other major structural brain disease
* Delirium within 30 days before the start of the screening period or a history of delirium
* At risk of suicide according to the Columbia-Suicide Severity Rating Scale (C-SSRS) (answers "yes" to Question 4 or 5 of the suicidal ideation section of the C-SSRS) or any suicide attempt within 6 months before the start of the screening period, or at serious risk of suicide in the opinion of the investigator or subinvestigator
* Prior or current treatment with anti-amyloid beta antibodies

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in CMAI score from baseline | up to week 12
  To assess agitation symptoms
Adverse events | up to week 16
  To Evaluate the Safety
Body weight | up to week 16
  To Evaluate the Safety
Body temperature | up to week 16
  To Evaluate the Safety
Blood pressure | up to week 16
  To Evaluate the Safety
Pulse rate | up to week 16
  To Evaluate the Safety
Respiratory rate | up to week 16
  To Evaluate the Safety
ECG RR interval | up to week 12
  To Evaluate the Safety
ECG PR interval | up to week 12
  To Evaluate the Safety
ECG QRS complex | up to week 12
  To Evaluate the Safety
ECG QT interval | up to week 12
  To Evaluate the Safety
ECG QTcF | up to week 12
  To Evaluate the Safety
Number of participants with abnormal laboratory tests (hematology) | up to week 12
  Hematology (PT, RBC count, RBC indices, WBC count, Differential, Hemoglobin, Hematocrit)
Number of participants with abnormal laboratory tests (Clinical chemistry) | up to week 12
  Clinical chemistry (Blood urea nitrogen (BUN), Potassium, Creatinine, Sodium, Glucose (fasting or nonfasting), Calcium, Chloride, Total protein, Albumin, Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Alkaline phosphatase, Total and direct bilirubin, Lactate dehydrogenase (LDH), Phospholipid, γ-Glutamyl transferase (GGT)
Number of participants with abnormal Blood coagulation profile (Activated partial thromboplastin time (APTT), Prothrombin time (PT), International normalized ratio (INR)) | up to week 12
  Blood coagulation (Activated partial thromboplastin time (APTT), Prothrombin time (PT), International normalized ratio (INR))
Number of participants with abnormal Urinalysis | up to week 12
  Urinalysis (pH, Glucose, Protein, Blood, Ketones)
COLUMBIA-SUICIDE SEVERITY RATING SCALE（C-SSRS） | up to week 16
  To Evaluate the Safety

SECONDARY OUTCOMES:
Cohen-Mansfield Agitation Inventory (CMAI) score at each visit and change from baseline | up to 12 week
  To Evaluate the Efficacy The range of CMAI score is 29-203. Higher score means a worse outcome.
Clinical Global Impression-Severity （CGI-S） score at each visit and change from baseline | up to 12 week
  To Evaluate the Efficacy The range of CGI-S score is 0-7. Higher score means a worse outcome.
Clinical Global Impression-Severity （CGI-S） score at each visit | up to 12 week
  To Evaluate the Efficacy
Neuropsychiatric Inventory in Nursing Home Version（NPI-NH） score at each visit and change from baseline | up to 12 week
  To Evaluate the Efficacy The range of NPI-NH score is 0-170. Higher score means a worse outcome.
Mini Mental State Exam(MMSE) score at baseline and Week 12, and change from baseline | up to 12 week
  To Evaluate the Efficacy The range of MMSE score is 0-30. Higher score means a better outcome.
Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL)score at baseline and Week 12, and change from baseline | up to 12 week
  To Evaluate the Efficacy The range of ADCS-ADL score is 0-78. Higher score means a better outcome.
Duration of the investigational medicinal product administration | up to 12 week
  To Evaluate the Efficacy
Pharmacokinetic assessments | up to 12 week
  Plasma ONO-2020 concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (38):
- Japan (38):
  - Hotei Hospital, Aichi
  - Akita Prefectural Center For Rehabilitation and Psychiatric Medicine, Akita
  - Medical Corporation Keishinkai Kyowa Hospital, Akita
  - Aiseikai General Incorporated Foundation, Hirosaki Aiseikai Hospital, Aomori
  - Seinan Hospital, Aomori
  - Fukui Hospital, Fukui
  - Matsubara Hospital, Fukui
  - Aburayama Hospital, Fukuoka
  - Kuramitsu Hospital, Fukuoka
  - Kishikai Kishi Hospital, Gunma
  - Hayakawa Clinic, Hiroshima
  - Koseikai Cocoro Hospital Kusatsu, Hiroshima
  - Nakamura Hospital, Hiroshima
  - Keiseikai Hospital, Hokkaido
  - NHO Obihiro National Hospital, Hokkaido
  - Airanomori Hospital, Kagoshima
  - Ishiki Hospital, Kagoshima
  - Sansyu Hospital, Kagoshima
  - Taniyama Hospital, Kagoshima
  - Fujisawahospital, Kanagawa
  - Hatano Kousei Hospital, Kanagawa
  - Showa Medical University Northern Yokohama Hospital, Kanagawa
  - Hosogi Hospital, Kochi
  - Ichiyo Mental Hospital, Kochi
  - Maizuru Medical Center, Kyoto
  - Nishiyama Hospital, Kyoto
  - Iryohojin Shadan Shoshinkai Morinohosupitaru・Aoba, Miyagi
  - JA-Nagano North Alps Medical Center Azumi Hospital, Nagano
  - Jizenkai Ando Hospital, Nagano
  - Nara Medical University Hospital, Nara
  - Nagaokai Neyagawa Sanatorium, Osaka
  - Osaka Institute of Clinical Psychiatry Shin-Abuyama Hospital, Osaka
  - Hizen Psychiatric Center, Saga
  - Rainbow & Sea Hospital, Saga
  - Saitama Konan Hospital, Saitama
  - Asuka Hospital, Tokyo
  - Nishigahara Hospital, Tokyo
  - Sanyokai Sanyo Hospital, Yamagata

IPD SHARING:
Plan to Share IPD: No